CLINICAL TRIAL: NCT01545700
Title: Effect of Low-Dose Dexamethasone on the Incidence of Hyperglycemia Following Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director, Cardiac Anesthesia and Clinical Research, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH08-413
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Complications
Keywords: dexamethasone; hyperglycemia; gynecologic surgery
MeSH Terms: conditions — Postoperative Complications; Hyperglycemia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Control, saline 0-4 hours (Placebo Comparator): 2 cc of saline
  Interventions: Drug: Control-saline
- Dexamethasone 4 mg, 0-4 hours (Active Comparator): Dexamethasone 4 mg administered intraoperatively
  Interventions: Drug: Dexamethasone 4 mg
- Dexamethasone 8 mg, 0-4 hours (Active Comparator): Dexamethasone 8 mg administered intraoperatively
  Interventions: Drug: Dexamethasone 8 mg
- Placebo Comparator saline 8-24 hours (Placebo Comparator): placebo, 2 cc saline
  Interventions: Drug: Control saline
- Dexamethasone 4 mg, 8-24 hours (Active Comparator): Dexamethasone 4 mg administered intraoperatively
  Interventions: Drug: Dexamethasone 4 mg
- Dexamethasone 8 mg, 8-24 hours (Active Comparator): Dexamethasone 8 mg administered intraoperatively
  Interventions: Drug: Dexamethasone 8 mg

INTERVENTIONS:
Drug: Control-saline — Patients are randomized to receive saline 2 cc
  Arms: Control, saline 0-4 hours
Drug: Dexamethasone 4 mg — Patients randomized to receive dexamethasone 4mg and 1 cc saline
  Arms: Dexamethasone 4 mg, 0-4 hours
Drug: Dexamethasone 8 mg — Patients randomized to receive dexamethasone 8mg
  Arms: Dexamethasone 8 mg, 0-4 hours
Drug: Control saline — Patients are randomized to receive saline 2 cc
  Arms: Placebo Comparator saline 8-24 hours
Drug: Dexamethasone 4 mg — Patients are randomized to receive dexamethasone 4 mg and saline 1 cc
  Arms: Dexamethasone 4 mg, 8-24 hours
Drug: Dexamethasone 8 mg — Patients are randomized to receive dexamethasone 8 mg
  Arms: Dexamethasone 8 mg, 8-24 hours

SUMMARY:
The question of a possible hyperglycemic effect from single-dose dexamethasone is an important issue for clinicians managing patients in the intraoperative and postoperative periods. Recent evidence suggests that even moderate elevations in blood glucose levels may be associated with adverse events.

The aim of this clinical investigation is to determine whether standard clinical doses of dexamethasone produce hyperglycemia in the perioperative period.

DETAILED DESCRIPTION:
Patients will be randomized on the morning of surgery to one of six groups; dexamethasone 4mg groups (0-4 hour group, 8-24 hour group), dexamethasone 8 mg groups (0-4 hour group, 8-24 hour group), or a placebo group(0-4 hour group, 8-24 hour group). Randomization will be performed using the sealed envelope method (on the basis of a block-randomized computer-generated list). The drug/placebo solution will be prepared by the pharmacy into a syringe (either 2cc of dexamethasone (8mg), 1cc dexamethasone (4mg) + 1cc normal saline, or 2cc of saline (placebo)) and delivered to one of investigators. All solutions are clear and appear identical. Patients in the dexamethasone groups will receive a standard intraoperative dose of dexamethasone (either 4mg or 8 mg) intravenously at the induction of anesthesia. Patients in the placebo groups will receive 2 cc of saline at induction of anesthesia. Study syringes will be prepared by the pharmacy, and all clinicians will be blinded to group assignment.

Primary Outcome Variable Serum Glucose levels: In the 0-4 hour patients, Blood glucose concentrations will be measured at 5 time intervals: at induction of anesthesia and at 60, 120, 180, and 240 minutes after the dexamethasone is administered. In the 8-24 hour patients, blood glucose levels will be measured at induction of anesthesia and at at 8- and 24-hours after induction. All blood samples will be measured using a portable glucometer which is calibrated daily. Blood glucose will be calculated by measuring a fingerprick capillary blood sample. The blood samples will be collected while the patient is under anesthesia and recovering from surgery.

Secondary Outcome Variables

1. Pain scores: Postoperative pain scores will be assessed using 100 mm visual analog scale (VAS) in which 0 represents no pain and 100 represents the worst pain imaginable. Pain scores will be measured at rest and with movement at 1 and 2 hours following surgery.
2. Nausea and vomiting scores: The incidence of nausea will be quantified using a verbal rating scale (VRS- 0=no nausea, 1=mild nausea, 2=moderate nausea, 3=severe nausea). The incidence of vomiting was quantified on a 4-point scale; 0 = (none) no episodes, 1= (mild) 1 episode, 2= (moderate) 2-3 episodes, 3= (severe) more than 3 episodes. Nausea and vomiting scores will be obtained at discharge from the PACU.
3. PACU data: Episodes of nausea and vomiting will be recorded. Requirements for pain medication and antiemetic medication will be recorded. The time needed to meet discharge criteria and achieve actual discharge will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for elective gynecologic surgery

Exclusion Criteria:

* Age < 18 or > 90, patients receiving chronic or preoperative steroids,or allergy to dexamethasone.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at NorthShore University HealthSystem (a single tertiary medical center affiliated with the University of Chicago Pritzker School of Medicine) and was registered with ClinicalTrials.gov (NCT #01545700). Participants were recruited by reviewing operating room schedules and contact by telephone on the day before surgery.
Pre-assignment Details: A total of 200 patients were enrolled in this clinical trial.
Groups:
- Control, Saline 0-4 Hours: 2 cc of saline
  Control-saline : Patients are randomized to receive saline 2 cc
- Dexamethasone 4 mg, 0-4 Hours: Dexamethasone 4 mg administered intraoperatively
  Dexamethasone 4 mg : Patients randomized to receive dexamethasone 4mg and 1 cc saline
- Dexamethasone 8 mg, 0-4 Hours: Dexamethasone 8 mg administered intraoperatively
  Dexamethasone 8 mg : Patients randomized to receive dexamethasone 8mg
- Placebo Comparator Saline 8-24 Hours: placebo, 2 cc saline
  Control saline : Patients are randomized to receive saline 2 cc
- Dexamethasone 4 mg, 8-24 Hours: Dexamethasone 4 mg administered intraoperatively
  Dexamethasone 4 mg : Patients are randomized to receive dexamethasone 4 mg and saline 1 cc
- Dexamethasone 8 mg, 8-24 Hours: Dexamethasone 8 mg administered intraoperatively
  Dexamethasone 8 mg : Patients are randomized to receive dexamethasone 8 mg
Period: Overall Study
Arm/Group | Control, Saline 0-4 Hours | Dexamethasone 4 mg, 0-4 Hours | Dexamethasone 8 mg, 0-4 Hours | Placebo Comparator Saline 8-24 Hours | Dexamethasone 4 mg, 8-24 Hours | Dexamethasone 8 mg, 8-24 Hours
Started | 34 | 33 | 33 | 34 | 33 | 33
Completed | 33 | 32 | 31 | 34 | 32 | 33
Not Completed | 1 | 1 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control, Saline 0-4 Hours | Dexamethasone 4 mg, 0-4 Hours | Dexamethasone 8 mg, 0-4 Hours | Placebo Comparator Saline 8-24 Hours | Dexamethasone 4 mg, 8-24 Hours | Dexamethasone 8 mg, 8-24 Hours | Total
Number analyzed (Participants) | 34 | 33 | 33 | 34 | 33 | 33 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 30 | 25 | 28 | 28 | 169
  >=65 years | 5 | 4 | 3 | 9 | 5 | 5 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10) | 53 (9) | 53 (11) | 57 (12) | 53 (13) | 56 (11) | 54 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 33 | 34 | 33 | 33 | 200
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 33 | 34 | 33 | 33 | 200

OUTCOME MEASURES:

1. Secondary Outcome: Pain Scores
Description: VAS pain scoes at rest 0=no pain, 100=worst pain imaginable
Time Frame: Patients were followed for the duration of hospitalization, for an average of 6 days
Measure: Mean (Standard Deviation); unit: 0-100 VAS scale scores on a scale
Groups:
- Placebo 0-4 Hours: Placebo 0-4 hours baseline
Arm/Group | Placebo 0-4 Hours | Dexamethasone 4 mg 0-4 Hours | Dexamethasone 8 mg 0-4 Hours | Placebo 8-24 Hours | Dexamethasone 4 mg 8-24 Hours | Dexamethasone 8 mg 8-24 Hours
Number analyzed (Participants) | 33 | 32 | 31 | 34 | 32 | 33
0-100 VAS scale scores on a scale | 50 (21) | 47 (26) | 45 (24) | 50 (21) | 45 (17) | 44.5 (23)

2. Primary Outcome: Serum Blood Glucose Concentrations
Description: Serum blood glucose concentrations
Time Frame: Patient were followed for the duration of hospitalization, for an average of 6 days
Population: per protocol
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Placebo 0-4 Hours-baseline: Placebo 0-4 hours baseline
- Placebo 0-4 Hours-1 Hour: Placebo 0-4 hours-1 hour
- Placebo 0-4 Hours-2 Hours: Placebo 0-4 hours-2 hours
Arm/Group | Placebo 0-4 Hours-baseline | Placebo 0-4 Hours-1 Hour | Placebo 0-4 Hours-2 Hours | Placebo 0-4 Hours-3 Hours | Placebo 0-4 Hours-4 Hours | Dexamethasone 4 mg 0-4 Hours-baseline | Dexamethasone 4 mg 0-4 Hours-1 Hour | Dexamethasone 4 mg 0-4 Hours-2 Hours | Dexamethasone 4 mg 0-4 Hours-3 Hours | Dexamethasone 4 mg 0-4 Hours-4 Hours | Dexamethasone 8 mg 0-4 Hours-baseline | Dexamethasone 8 mg 0-4 Hours-1 Hour | Dexamethasone 8 mg 0-4 Hours-2 Hours | Dexamethasone 8 mg 0-4 Hours-3 Hours | Dexamethasone 8 mg 0-4 Hours-4 Hours | Placebo 8-24 Hours Baseline | Placebo 8-24 Hours-8 Hours | Placebo 8-24 Hours-24 Hours | Dexamethasone 4 mg 8-24 Hours-baseline | Dexamethasone 4 mg 8-24 Hours-8 Hours | Dexamethasone 4 mg 8-24 Hours-24 Hours | Dexamethasone 8 mg 8-24 Hours-baseline | Dexamethasone 8 mg 8-24 Hours-8 Hours | Dexamethasone 8 mg 8-24 Hours-24 Hours
Number analyzed (Participants) | 34 | 33 | 33 | 33 | 33 | 32 | 32 | 32 | 32 | 32 | 31 | 31 | 31 | 31 | 31 | 34 | 34 | 34 | 32 | 32 | 32 | 33 | 33 | 33
mg/dl | 101 (15) | 137 (29) | 140 (28) | 141 (34) | 139 (34) | 107 (21) | 141 (23) | 159 (33) | 159 (30) | 159 (25) | 108 (23) | 138 (27) | 151 (23) | 146 (22) | 149 (25) | 101 (19) | 150 (36) | 121 (26) | 98 (16) | 149 (28) | 119 (16) | 100 (19) | 151 (36) | 124 (27)

ADVERSE EVENTS:
Groups:
- Dexamethasone Group: either 4 mg or 8 mg
Arm/Group | Control-saline Group | Dexamethasone Group
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/128
Other Adverse Events (participants affected / at risk) | 0/67 | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes